CLINICAL TRIAL: NCT04957407
Title: The Research of Constructing a Risk Assessment Model for Gastric Cancer Based on Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 71804161
Record Dates: First submitted 2021-07-08; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Gastric Cancer; Precancerous Lesion; Mechine Learning
MeSH Terms: conditions — Stomach Neoplasms | interventions — Pepsinogen A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- non-atrophic gastritis: OLGA-0 group；OLGA (Operative Link on Gastritis Assessment)
- mild-moderate atrophic gastritis: OLGA I-II group；OLGA (Operative Link on Gastritis Assessment)
- severe atrophic gastritis: OLGA III-IV group；OLGA (Operative Link on Gastritis Assessment)
  Interventions: Other: pepsinogen
- gastric cancer: gastric cancer
  Interventions: Other: pepsinogen

INTERVENTIONS:
Other: pepsinogen — diagnostic value of pepsinogen for severe atrophy and gastric cancer
  Groups: gastric cancer; severe atrophic gastritis

SUMMARY:
Based on the gastric cancer database established earlier, this project explored the PG standard suitable for Chinese people, and further explored the establishment of machine learning model to stratify gastric cancer risk in the population, guide the frequency of gastroscopy screening, and extract important gastric cancer risk factors from it.Establish electronic health records of gastric organs, track the development and outcome of gastric diseases through deep learning method, in order to predict the development and outcome of gastric diseases;Then, the simulation hypothesis deductive method is used to compare the outcomes that may be caused by different lifestyles with the help of deep learning model, so as to guide patients to develop a better lifestyle and explore the establishment of health management paths for gastric cancer patients and high-risk groups in China.

ELIGIBILITY:
Inclusion Criteria:

* 1） intention to undergo gastroscopy during health checkup examination; and 2) 25-75 years of age

Exclusion Criteria:

* 1) a history of gastric ulcer, gastric polyp, or GC; 2) a history of gastrectomy; 3) treatment with a proton pump inhibitor in the last month; 4) contraindications to gastroscopy; 5) a history of Hp eradication; 6) a history of abdominal pain, abdominal distention, belching, acid reflux, nausea and other digestive tract symptoms within 1 month or 67) incomplete data.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive subjects who underwent regular health checkup at nine International Healthcare
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
pepsinogen value for precanceous lesion and Gastric cancer | 1 year
  pepsinogen value for precanceous lesion and Gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yuling Tong, Dr., Principal Investigator — 2nd affiliated hospital of Zhejiang University, school of medicine
Locations (2):
- China (2):
  - Zhejiang Provincial Hospital of Traditional Chinese Medicine, Hangzhou
  - Ningbo cadres health center, Ningbo